CLINICAL TRIAL: NCT03328663
Title: Randomized Trial of a Psychological Intervention to Promote Coping for Caregivers of Patients Undergoing Hematopoietic Stem Cell Transplantation (HCT)
Brief Title: Psychological Intervention for Caregivers of Patients Undergoing Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-476; CA087723 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: Cancer Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CARE intervention (Experimental): * Six psychological intervention sessions in-person or via video conferencing conducted by a trained psychologist
  * The CARE intervention contain 3 component
    * a psychoeducational component to address preparednessmanage expectations, and develop caregiving skills
    * a psychosocial component focusing on coping strategies, mindfulness, and facilitating acceptance while living with uncertainty
    * a self-care component to promote caregiver health and well-being
  Interventions: Other: CARE
- Standard transplant care (Active Comparator): * Standard Transplant Care
  * Social work consults to help caregivers only upon request
  Interventions: Other: CARE; Other: Standard Transplant Care

INTERVENTIONS:
Other: CARE — Promote effective coping and reduce caregiving burden.
Other: Standard Transplant Care — Standard cared administered by the hospital.
  Arms: Standard transplant care

SUMMARY:
This research study is evaluating the impact of a psychological intervention on the quality of life and mood of caregivers of patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
The purpose of this study is to find out whether a psychological intervention can make the experience of being a caregiver more manageable by improving the participant's quality of life, mood, and caregiving burden during the participant's loved one's transplant process.

The psychological intervention will entail six visits with a trained clinician and will take place during the first three months of the participant's loved ones' transplant process. A trained behavioral psychologist or social worker will meet with the participant or talk with the participant over the telephone or video conference for 45 minutes at a time to discuss the participant's caregiver experience and to help the participant develop effective skills to support the participant's loved one as well as participant over the course of the transplant.

The study will use a series of questionnaires to measure the participant's quality of life, mood, and overall caregiving burden. Study questionnaires will be completed in the hospital or clinic. The participant will also have the option of completing these questionnaires remotely through a secure web link, over the telephone, or in a mailed paper copy.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers (≥18 years) of patients undergoing autologous or allogeneic HCT at MGH, and they must attend the HCT consent visit with the patient.
* A relative or a friend who either lives with the patient or has in-person contact with him or her at least twice per week and is identified as the primary caregiver for transplant.
* Ability to speak English or able to complete questionnaires with minimum assistance of an interpreter.

Exclusion Criteria:

• Significant uncontrolled psychiatric or other co-morbid disease, which the primary oncologist believes prohibits the ability to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention (feasibility description below) | 2 years
  Feasibility defined if at least 60% of eligible caregivers are enrolled in the study and attend at least 50% of the intervention visits

SECONDARY OUTCOMES:
Compare Caregiver QOL (CarGOQOL) between the study arms | up to day +90
  we will compare caregiver QOL as measured by CarGOQOL at day +30 and day +90 after the intervention (adjusting for baseline values)
Compare caregiving burden (CRA) between the study arms | up to day +90
  we will compare caregiver caregiving burden as measured by Caregiver Reaction Assessment (CRA) at day +30 and day +90 after the intervention (adjusting for baseline values)
Compare caregiver mood (HADS) between the study arms | up to day +90
  We will compare caregiver mood use the Hospital Anxiety and Depression Scale (HADS) at day +30 and day +90 (controlling for baseline values). The HADS includes two subscales: depression (range 0 (no distress) to 21 (maximum distress) and anxiety (range 0 (no distress) and 21 (maximum distress))
Compare caregiver self-efficacy (CASE-t) between the study arms | up to day +90
  We will compare caregiver self-efficacy using the Cancer Self-Efficacy Scale-transplant (CASE-t) at day +30 and day +90 (controlling for baseline values). The scale ranges from 0 to 170 with higher scores indicate higher self efficacy
Compare perceived coping skills (MOCS) between the study arms | up to day +90
  Compare caregiver coping skills using the Measure of Current Status (MOCS) between the study arms. Score ranges from 0-52, with higher scores indicating higher coping skills

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No